CLINICAL TRIAL: NCT06634771
Title: Frontal E/I Balance Mediation of TACS Effects on Behavioral Flexibility
Brief Title: Flexibility, Alcohol Misuse, and Excitation
Acronym: FLAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Charlotte Boettiger, PhD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23-1702; P60AA011605 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Behavioral Flexibility; Healthy Volunteers; High Risk Alcohol Use
Keywords: alcohol; brain stimulation; MRI; EEG

STUDY DESIGN:
Intervention Model Description: Study design consists of 3 groups of participants:
  1. Control (CON): no adolescent binge drinking (AIE) and current (past month) World Health Organization (WHO) risk drinking levels of either 0 or 1 (abstinent or low-risk)
  2. (RISK): no AIE and current WHO level 2, 3, or 4 (medium risk, high risk, or very high risk)
  3. (RISK+AIE): history of adolescent binge drinking and current WHO risk level 2, 3, or 4.
  Within each group (n=22), participants will be randomly assigned to either the 10Hz tACS (stim) group or the sham tACS (sham) group.
  Study design requires randomly assigning individuals to a stimulation group after completing Session 1. Prior to study onset, Dr. Boettiger will create a randomization table in which stimulation type (true or sham) is pseudo randomly ordered within groups, stratified by sex. Dr. Boettiger will provide assignment to the study team based on this predefined randomization table in order to ensure balanced sex and group for each stimulation type.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study team will be provided a numeric code to enter into the XCSITE 100 tACS system, which will conceal the stimulation parameters from the study team, ensuring double blinding. The XSCITE 100 device allows for the programming of stimulation codes corresponding to sham or active stimulation, both of which are set to a total duration of 30 minutes, allowing for reliable double-blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10Hz bi-frontal tACS (Experimental): For Session 3, participants will complete a Habitual Association between Images Task (HABIT) Test Session in the Howell Hall Neurostimulation Core Lab or electroencephalogram (EEG) Core Lab, which is located one floor below the Boettiger Lab. Participants will receive either 10Hz bi-frontal transcranial alternating current stimulation (tACS) or sham tACS.
  10 Hz bi-frontal tACS: Alternating current stimulation is delivered by an XCSITE 100 device (Pulvinar Neuro, Chapel Hill, NC), through three conductive carbon-rubber electrodes. Electrodes are placed over the apex of the head (Cz) and the prefrontal cortex bilaterally (F3 and F4). Stimulation is delivered during the second half of the HABIT Test session. Stimulation parameters: 2mA peak-to-peak 10Hz sine-wave flanked by 10 second linear envelope ramps in and out for a total duration of 30 min and 20 seconds.
  Interventions: Device: 10 Hz transcranial alternating current stimulation (tACS)
- sham tACS (Sham Comparator): Sham transcranial alternating current stimulation (tACS): The procedure for sham stimulation will be identical, but the actual stimulation will last for 2 minutes instead of 30 minutes. Participants generally report that stimulation is felt most strongly at the beginning of active stimulation, before they adjust to the sensation. Sham stimulation is meant to mimic this progression in terms of tactile salience. Stimulation is delivered for 2 minutes at the beginning of the HABIT reversal task, flanked by 10 second linear envelope ramps. The stimulating electrodes are left on the head until completion of the HABIT task, as is the case in active stimulation. There is no visual or auditory indication to the participant or researcher when the 2-minute sham stimulation period has ended, allowing the sham stimulation condition to feel similar to active stimulation.
  Interventions: Device: sham transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: 10 Hz transcranial alternating current stimulation (tACS) — 10 Hz bi-frontal tACS: Alternating current stimulation is delivered by an XCSITE 100 device (Pulvinar Neuro, Chapel Hill, NC), through three conductive carbon-rubber electrodes. Electrodes are placed over the apex of the head (Cz) and the prefrontal cortex bilaterally (F3 and F4). Stimulation is delivered during the second half of the HABIT Test session. Stimulation parameters: 2mA peak-to-peak 10Hz sine-wave flanked by 10 second linear envelope ramps in and out for a total duration of 30 min and 20 seconds.
  Arms: 10Hz bi-frontal tACS
Device: sham transcranial alternating current stimulation (tACS) — Sham tACS: The procedure for sham stimulation will be identical, but it will last for 2 minutes instead of 30 minutes.
  Arms: sham tACS

SUMMARY:
The goal of this study is to learn whether a single non-invasive brain stimulation alpha-transcranial alternating current stimulation (alpha-tACS) session changes measures of excitability in the prefrontal cortex. It will also learn whether these changes predict differences in habitual action selection in a laboratory task and whether the effects depend on alcohol use history. The main questions it aims to answer are:

Does alpha-tACS reduce habitual action selection by reducing excitability in the prefrontal cortex? Is alpha-tACS most effective in reducing habitual action selection in hazardous drinkers who engaged in binge-drinking during adolescence?

Researchers will compare alpha-tACS to sham stimulation to see if alpha-tACS changes habitual action selection by changing prefrontal excitability.

Participants will:

Visit the lab for behavioral training Visit the imaging center for an MRI session Visit the lab to receive alpha-tACS or sham stimulation during behavioral testing and undergo EEG recordings before and after stimulation Visit the imaging center for a repeat MRI session Provide a small sample of blood from a finger-prick in the first and last visits.

DETAILED DESCRIPTION:
This study is designed to probe the role of the balance between excitatory (E) and inhibitory (I) signaling (E/I) in key nodes of control circuitry in mediating the relationship between alcohol misuse and inflexible behavior. In addition, the investigators aim to determine whether adolescent binge alcohol exposure amplifies the effects of binge exposure in adulthood. The investigators will accomplish this goal via a single multi-session study. Participants (n=66) will comprise three groups: adults self-reporting high risk drinking [World Health Organization (WHO) risk levels 2, 3, or 4], with (n=22) or without (n=22) a history of adolescent alcohol misuse (AIE), and lifetime low risk drinking adults (WHO risk levels 0 or 1; n=22).

Design: a 3-session study that includes an initial screening session and behavioral training (Session 1), behavioral testing and a magnetic resonance imaging (MRI) scan session (Session 2), bifrontal 10Hz-transcranial alternating current stimulation (tACS; true or sham) during behavioral testing with pre- and post-electroencephalogram (EEG) recording in a resting-state, followed by a second MRI scan session (Session 3). The investigators predict that adolescent and adult binge history will have interacting effects on E/I balance indices derived from EEG and magnetic resonance spectroscopy (MRS) and on behavioral flexibility measured in the Hidden Association between Images Task (HABIT) Test and that E/I balance indices will mediate the relationship between alcohol misuse and behavioral flexibility. The investigators also propose to test a causal relationship between E/I balance and behavioral flexibility by testing whether 10Hz-tACS to bilateral dorsolateral prefrontal cortex (dlPFC) alters habitual action selection in the HABIT Test in proportion to its effects on the dlPFC 1/f EEG slope and/or the MRS-derived gamma-amino-butyric acid (GABA)/glutamate+glutamine (Glx) ratio. The investigators predict that changes in indices of E/I balance induced by tACS will inversely associate with changes in habitual response selection. The investigators will collect a small amount of blood from a finger prick in Sessions 1 and 3 will use the collected dried blood spots to measure inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* • 22-50 years old

  * Have a high school diploma or equivalent
  * Medically healthy
  * Fluent in English

For RISK group only:

* High risk alcohol use in the past month [World Health Organization (WHO ) risk level 2-4]
* No history of adolescent binge drinking

For RISK+ Adolescent binge alcohol (AIE) group only:

* High risk alcohol use in the past month (WHO risk level 2-4)
* High levels of adolescent alcohol use (4 or more binge drinking episodes before age 18)

For Control (CON) group only:

* Low risk alcohol use throughout the lifetime (WHO risk level 0-1)
* No history of adolescent binge drinking
* No lifetime history of Alcohol Use Disorder (AUD)

Exclusion Criteria:

* Any individual who meets one or more of the following criteria will be excluded from participation [excluding positive breath alcohol concentration (BAC), urine drug screen, psychiatric diagnoses, and color blindness, all will be self-reported]:

  * Lifetime history of a substance use disorder (SUD; including nicotine) but participants will not be excluded for an AUD.
  * Neurological disease such as dementia, seizures or head trauma
  * History of psychosis or psychotic episodes
  * Diagnosis of attention deficit hyperactivity disorder (ADHD)
  * Any systemic or inflammatory disease that could affect cognitive functioning (e.g., cancer, cardiovascular disease)
  * Any motor or visual disturbances that could hinder task performance (e.g., color blindness)
  * Use of psychoactive recreational drugs in the past month (excluding caffeine and alcohol)
  * Use of psychotropic medications in the past month including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics (excluding antidepressant use when dosage has been stable for 1 month or longer)
  * Use of therapeutic brain stimulation [e.g. transcranial magnetic stimulation (TMS) or electroconvulsive therapy (ECT)] in the past month
  * Any history of brain surgery
  * History of migraine headaches
  * Pregnancy
  * Any brain implants or devices
  * First degree relative with primary epilepsy
  * Claustrophobia
  * Any magnetic resonance imaging (MRI) contraindication based on the University of North Carolina Biomedical Research Imaging Center's MRI safety checklist
  * Breath alcohol above 0.0% at time of session
  * Positive urine drug screen at time of session

If a participant should have an exclusion criterion arise in the course of their participation (e.g. pregnancy or psychotic episode), their participation in the study will end unless the circumstances are transitory in nature (e.g. positive breath alcohol or urine drug screen).

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in habitual action selection | at study completion, an average of 2 weeks
  Habitual action selection is calculated as the proportion of perseverative errors after Stimulus-Response contingency change for highly trained (Familiar) stimuli in the Hidden Association between Images Task (HABIT). The researchers will compare habitual responding pre- and post-transcranial alternating current stimulation (tACS).
Prefrontal GABA:glutamate/glutamine ratio | at study completion, an average of 2 weeks
  The researchers will evaluate the difference in these ratios measured via single voxel magnetic resonance spectroscopy (MRS). These data will be used to compare groups as well as to assess the correlation between these ratios and behavioral flexibility and alcohol misuse measures.

SECONDARY OUTCOMES:
Inflammatory markers | at study completion, an average of 2 weeks
  The researchers will measure the effect of transcranial alternating current stimulation (tACS) of bilateral dorsolateral prefrontal cortex on circulating inflammatory markers, including C-reactive protein, interleukin -6 (IL-6), and tumor necrosis factor-alpha (TNF-alpha). These data will also be used to assess the correlation between these markers and behavioral flexibility and alcohol misuse measures.
Control circuit functional connectivity | at study completion, an average of 2 weeks
  The effect of 10Hz-tACS on resting-state functional connectivity (FC) of the dlPFC and the aIC with other brain regions of interest, as well as whole brain analyses. FC will be used as the mediating variable, change in HABIT perseverative errors will serve as the dependent variable and will be adjusted for sex, age, education, baseline perseverative error, and psychiatric diagnoses; tACS group will serve as the independent variable; AIE and current alcohol misuse scores will serve as moderating variables.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte A Boettiger, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Brief summary of the assessment schedule for data that will eventually be shared with the NIAAADA:
  In this 3-visit study, eligibility is first determined at the screening and randomization visit; dried blood spot measures of inflammatory markers will also be collected. In visit 2, measures of baseline habitual action selection in the HABIT, structural MRI, baseline resting-state fMRI, and single-voxel MRS measuring GABA and glutatmate/glutamine will be collected. At visit 3, resting-state EEG before and after 10Hz- or sham-tACS, as well as habitual action selection in the HABIT during 10Hz- or sham-tACS, as well as repeat structural and functional MRI and MRS, and dried blood spot collection following 10Hz- or sham-tACS will be collected. Demographic, psychometric, and substance-related information will be collected via REDCap at the participant's convenience. Data will be uploaded to the PI's NIMH Data Archive (NDA) account by established deadlines.
Supporting Information: SAP
Time Frame: Upon approval of the study data structure by the NIMH Data Archive (NDA), data will be uploaded every six months.
  For each manuscript based on findings from this project, investigators will submit to the NDA: data, list of variables, analytic plan, and results.
Access Criteria: The researchers will determine who will have access to which aspects of the project data based on NIH's data access principles. The researchers will provide access to person-level data for research purposes only, based on Data Use Certifications. Data on UNC servers will be made available to investigators with appropriate IRB approval and Data Use Agreements.
URL: https://nda.nih.gov/niaaa

REFERENCES:
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- [Background] Wood W, Runger D. Psychology of Habit. Annu Rev Psychol. 2016;67:289-314. doi: 10.1146/annurev-psych-122414-033417. Epub 2015 Sep 10. PMID 26361052
- [Background] Viner RM, Taylor B. Adult outcomes of binge drinking in adolescence: findings from a UK national birth cohort. J Epidemiol Community Health. 2007 Oct;61(10):902-7. doi: 10.1136/jech.2005.038117. PMID 17873228
- [Background] Vanderhasselt MA, De Raedt R, Brunoni AR, Campanha C, Baeken C, Remue J, Boggio PS. tDCS over the left prefrontal cortex enhances cognitive control for positive affective stimuli. PLoS One. 2013 May 21;8(5):e62219. doi: 10.1371/journal.pone.0062219. Print 2013. PMID 23704874
- [Background] Smittenaar P, FitzGerald TH, Romei V, Wright ND, Dolan RJ. Disruption of dorsolateral prefrontal cortex decreases model-based in favor of model-free control in humans. Neuron. 2013 Nov 20;80(4):914-9. doi: 10.1016/j.neuron.2013.08.009. Epub 2013 Oct 24. PMID 24206669
- [Background] Siqueira L, Smith VC; COMMITTEE ON SUBSTANCE ABUSE. Binge Drinking. Pediatrics. 2015 Sep;136(3):e718-26. doi: 10.1542/peds.2015-2337. PMID 26324872
- [Background] Sellers KK, Mellin JM, Lustenberger CM, Boyle MR, Lee WH, Peterchev AV, Frohlich F. Transcranial direct current stimulation (tDCS) of frontal cortex decreases performance on the WAIS-IV intelligence test. Behav Brain Res. 2015 Sep 1;290:32-44. doi: 10.1016/j.bbr.2015.04.031. Epub 2015 Apr 28. PMID 25934490
- [Background] Rehm J, Shield KD, Roerecke M, Gmel G. Modelling the impact of alcohol consumption on cardiovascular disease mortality for comparative risk assessments: an overview. BMC Public Health. 2016 Apr 28;16:363. doi: 10.1186/s12889-016-3026-9. PMID 27121289
- [Background] Ostlund SB, Balleine BW. Lesions of medial prefrontal cortex disrupt the acquisition but not the expression of goal-directed learning. J Neurosci. 2005 Aug 24;25(34):7763-70. doi: 10.1523/JNEUROSCI.1921-05.2005. PMID 16120777
- [Background] Olsen RW, Liang J. Role of GABAA receptors in alcohol use disorders suggested by chronic intermittent ethanol (CIE) rodent model. Mol Brain. 2017 Sep 20;10(1):45. doi: 10.1186/s13041-017-0325-8. PMID 28931433
- [Background] Miller EK, Cohen JD. An integrative theory of prefrontal cortex function. Annu Rev Neurosci. 2001;24:167-202. doi: 10.1146/annurev.neuro.24.1.167. PMID 11283309
- [Background] McKim TH, Dove SJ, Robinson DL, Frohlich F, Boettiger CA. Addiction history moderates the effect of prefrontal 10-Hz transcranial alternating current stimulation on habitual action selection. J Neurophysiol. 2021 Mar 1;125(3):768-780. doi: 10.1152/jn.00180.2020. Epub 2020 Dec 23. PMID 33356905
- [Background] McKim TH, Bauer DJ, Boettiger CA. Addiction History Associates with the Propensity to Form Habits. J Cogn Neurosci. 2016 Jul;28(7):1024-38. doi: 10.1162/jocn_a_00953. Epub 2016 Mar 11. PMID 26967944
- [Background] Matsumoto H, Ugawa Y. Adverse events of tDCS and tACS: A review. Clin Neurophysiol Pract. 2016 Dec 21;2:19-25. doi: 10.1016/j.cnp.2016.12.003. eCollection 2017. PMID 30214966
- [Background] Lam NH, Borduqui T, Hallak J, Roque A, Anticevic A, Krystal JH, Wang XJ, Murray JD. Effects of Altered Excitation-Inhibition Balance on Decision Making in a Cortical Circuit Model. J Neurosci. 2022 Feb 9;42(6):1035-1053. doi: 10.1523/JNEUROSCI.1371-20.2021. Epub 2021 Dec 9. PMID 34887320
- [Background] Kearney-Ramos TE, Dowdle LT, Lench DH, Mithoefer OJ, Devries WH, George MS, Anton RF, Hanlon CA. Transdiagnostic Effects of Ventromedial Prefrontal Cortex Transcranial Magnetic Stimulation on Cue Reactivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jul;3(7):599-609. doi: 10.1016/j.bpsc.2018.03.016. Epub 2018 Apr 10. PMID 29776789
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Hasin DS, Stinson FS, Ogburn E, Grant BF. Prevalence, correlates, disability, and comorbidity of DSM-IV alcohol abuse and dependence in the United States: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2007 Jul;64(7):830-42. doi: 10.1001/archpsyc.64.7.830. PMID 17606817
- [Background] Guerri C, Pascual M. Mechanisms involved in the neurotoxic, cognitive, and neurobehavioral effects of alcohol consumption during adolescence. Alcohol. 2010 Feb;44(1):15-26. doi: 10.1016/j.alcohol.2009.10.003. PMID 20113871
- [Background] Grant BF, Goldstein RB, Saha TD, Chou SP, Jung J, Zhang H, Pickering RP, Ruan WJ, Smith SM, Huang B, Hasin DS. Epidemiology of DSM-5 Alcohol Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions III. JAMA Psychiatry. 2015 Aug;72(8):757-66. doi: 10.1001/jamapsychiatry.2015.0584. PMID 26039070
- [Background] Grant BF, Chou SP, Saha TD, Pickering RP, Kerridge BT, Ruan WJ, Huang B, Jung J, Zhang H, Fan A, Hasin DS. Prevalence of 12-Month Alcohol Use, High-Risk Drinking, and DSM-IV Alcohol Use Disorder in the United States, 2001-2002 to 2012-2013: Results From the National Epidemiologic Survey on Alcohol and Related Conditions. JAMA Psychiatry. 2017 Sep 1;74(9):911-923. doi: 10.1001/jamapsychiatry.2017.2161. PMID 28793133
- [Background] Gbadeyan O, McMahon K, Steinhauser M, Meinzer M. Stimulation of Dorsolateral Prefrontal Cortex Enhances Adaptive Cognitive Control: A High-Definition Transcranial Direct Current Stimulation Study. J Neurosci. 2016 Dec 14;36(50):12530-12536. doi: 10.1523/JNEUROSCI.2450-16.2016. PMID 27974612
- [Background] Friedman NP, Robbins TW. The role of prefrontal cortex in cognitive control and executive function. Neuropsychopharmacology. 2022 Jan;47(1):72-89. doi: 10.1038/s41386-021-01132-0. Epub 2021 Aug 18. PMID 34408280
- [Background] Ersche KD, Gillan CM, Jones PS, Williams GB, Ward LH, Luijten M, de Wit S, Sahakian BJ, Bullmore ET, Robbins TW. Carrots and sticks fail to change behavior in cocaine addiction. Science. 2016 Jun 17;352(6292):1468-71. doi: 10.1126/science.aaf3700. PMID 27313048
- [Background] Ewing SW, Sakhardande A, Blakemore SJ. The effect of alcohol consumption on the adolescent brain: A systematic review of MRI and fMRI studies of alcohol-using youth. Neuroimage Clin. 2014 Jul 5;5:420-37. doi: 10.1016/j.nicl.2014.06.011. eCollection 2014. PMID 26958467
- [Background] Degenhardt L, O'Loughlin C, Swift W, Romaniuk H, Carlin J, Coffey C, Hall W, Patton G. The persistence of adolescent binge drinking into adulthood: findings from a 15-year prospective cohort study. BMJ Open. 2013 Aug 19;3(8):e003015. doi: 10.1136/bmjopen-2013-003015. PMID 23959750
- [Background] Davies M. The role of GABAA receptors in mediating the effects of alcohol in the central nervous system. J Psychiatry Neurosci. 2003 Jul;28(4):263-74. PMID 12921221
- [Background] Crews FT, Vetreno RP, Broadwater MA, Robinson DL. Adolescent Alcohol Exposure Persistently Impacts Adult Neurobiology and Behavior. Pharmacol Rev. 2016 Oct;68(4):1074-1109. doi: 10.1124/pr.115.012138. PMID 27677720
- [Background] Cohen E, Feinn R, Arias A, Kranzler HR. Alcohol treatment utilization: findings from the National Epidemiologic Survey on Alcohol and Related Conditions. Drug Alcohol Depend. 2007 Jan 12;86(2-3):214-21. doi: 10.1016/j.drugalcdep.2006.06.008. Epub 2006 Aug 17. PMID 16919401
- [Background] Brunye TT, Elliott G, Loverro K. Examining state-dependent effects of transcranial direct current stimulation on visual search and executive function tasks. Neuroreport. 2021 Jan 6;32(1):1-7. doi: 10.1097/WNR.0000000000001549. PMID 33165194
- [Background] Brosnan MB, Wiegand I. The Dorsolateral Prefrontal Cortex, a Dynamic Cortical Area to Enhance Top-Down Attentional Control. J Neurosci. 2017 Mar 29;37(13):3445-3446. doi: 10.1523/JNEUROSCI.0136-17.2017. No abstract available. PMID 28356395
- [Background] Boettiger CA, D'Esposito M. Frontal networks for learning and executing arbitrary stimulus-response associations. J Neurosci. 2005 Mar 9;25(10):2723-32. doi: 10.1523/JNEUROSCI.3697-04.2005. PMID 15758182